CLINICAL TRIAL: NCT05791188
Title: Electrolyte Disorders in Prediabetics and in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa Saad, Doctor, Assiut University
Other Study IDs: Electrolytes Diabetes Mellitus
Record Dates: First submitted 2023-03-16; First posted 2023-03-30 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Type 2 Diabetes Mellitus and Electrolyte Disorders
Keywords: electrolytes diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1- Prediabetics: Prediabetics who will be diagnosed by:
  Glycated hemoglobin (HbA1C) test 5.7 - 6.4% % on two separate tests
  Fasting blood sugar test 110-125 mg/dL (6.1 - 6.9 mmol/L) on two separate tests.
  Glucose tolerance test 140 - 179 mg/dL (7.8 - 9.9 mmol/L)
- 2- Diabetic patients without complications: Patients with Type 2 diabetes who will be diagnosed by:
  Glycated hemoglobin (HbA1C) test ≥ 6.5% on two separate tests
  Fasting blood sugar test ≥ 126 mg/dL (7 mmol/L) on two separate tests
  Glucose tolerance test ≥ 200 mg/dL (11.1 mmol/L) Random blood sugar test ≥ 200 mg/dL (11.1 mmol/L)
- 3- Diabetic patients with complications: Diabetic patients with complications (nephropathy, neuropathy, cardiovascular, retinopathy, metabolic disorders, diabetic ketoacidosis)
- 4- Controls: apparently normal subjects who have matched age and sex with patients groups

SUMMARY:
The aim of the study is to assess serum sodium [Na+], potassium [K+] magnesium [Mg2+], calcium [Ca2+], and chloride [Cl-] levels in patients who are prediabetic, diabetics and diabetic with complications (Diabetes mellitus type 2)

DETAILED DESCRIPTION:
Diabetes mellitus is a chronic disease that imposes enormous socioeconomic burdens attributable to complications of various bodily systems. Diabetes affected 463 million people (9.3% of all people) in 2019 and will affect 700 million (10.9%) by 2045.

According to the International Diabetes Federation (IDF), the prevalence of diabetes mellitus among Egyptian adults is 15.2%, which may be an underestimation. Therefore, diabetes mellitus should be thoroughly explored in terms of its risk factors, prevention, treatment, and consequences. Moreover, the general population should be aware of and well informed about all aspects of diabetes.

Prediabetes is a precursor before the diagnosis of diabetes mellitus. Adults with prediabetes often may show no signs or symptoms of diabetes but will have blood glucose levels higher than normal. The normal blood glucose level is between 70 - 99 mg/dL. In patients with prediabetes, the blood glucose levels elevated between 110 - 125 mg/dL.

Once the patient is diagnosed as prediabetes, he should be checked for progression to type 2 diabetes every one to two years. So early detection of prediabetes and so lifestyle changes through improved nutrition and physical activity are the first line treatment for preventing the transition from prediabetes to diabetes which can be as high as 70%.

A normal HbA1C level is below 5.7%, a level of 5.7-6.4% indicates prediabetes, and a level of 6.5% or more indicates diabetes. Within the 5.7-6.4% prediabetes range, the higher HbA1C, the greater risk is for developing type 2 diabetes.

Serum electrolytes are important cofactors for multiple enzymes and play a pivotal role in many key biological and physiological processes, including glucose metabolism. The excess or deficiency of these electrolytes was found to be linked to deleterious metabolism status.

Diabetic patients frequently develop a constellation of electrolyte disorders. These disturbances are particularly common in decompensated diabetics, especially in the context of diabetic ketoacidosis or nonketotic hyperglycemic hyperosmolar syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prediabetes who will be diagnosed by:

  * Glycated hemoglobin (HbA1C) test (6.1 - 6.4%) on two separate tests
  * Fasting blood sugar test 110-125 mg/dL (5.6 - 6.9 mmol/L) on two separate tests.
  * Glucose tolerance test 140 - 179 mg/dL (7.8 - 9.9 mmol/L)
* Patients with Type 2 diabetes who will be diagnosed by:

  * Glycated hemoglobin (HbA1C) test ≥ 6.5% on two separate tests
  * Fasting blood sugar test ≥ 126 mg/dL (7 mmol/L) on two separate tests
  * Glucose tolerance test ≥ 200 mg/dL (11.1 mmol/L)
  * Random blood sugar test ≥ 200 mg/dL (11.1 mmol/L)
* Patients with diabetic complications (nephropathy, neuropathy, cardiovascular, retinopathy, metabolic disorders, diabetic ketoacidosis)

Exclusion Criteria:

• Patients with Type 1 diabetes

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Prediabetics
  Diabetic patients (type 2 diabetes mellitus) without complications
  Diabetic patients (type 2diabetes mellitus) with complications
  Controls
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Serum sodium | baseline
  assessment of serum sodium [Na+] in prediabetic and diabetic patients compared with controls
Serum potassium | baseline
  assessment of serum potassium [K+] in prediabetic and diabetic patients compared with controls
Serum magnesium | baseline
  assessment of serum magnesium [Mg2+] in prediabetic and diabetic patients compared with controls
Serum calcium | baseline
  assessment of serum calcium [Ca2+] in prediabetic and diabetic patients compared with controls
Serum chloride | baseline
  assessment of serum chloride [Cl-] in prediabetic and diabetic patients compared with controls

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Faisal El-Adawy, Lecturer, Study Director — Assiut University

REFERENCES:
- [Background] Choi JH, Kim HR, Song KH. Musculoskeletal complications in patients with diabetes mellitus. Korean J Intern Med. 2022 Nov;37(6):1099-1110. doi: 10.3904/kjim.2022.168. Epub 2022 Oct 27. PMID 36300322
- [Background] Abouzid MR, Ali K, Elkhawas I, Elshafei SM. An Overview of Diabetes Mellitus in Egypt and the Significance of Integrating Preventive Cardiology in Diabetes Management. Cureus. 2022 Jul 20;14(7):e27066. doi: 10.7759/cureus.27066. eCollection 2022 Jul. PMID 36000101
- [Background] Eshak ES, Iso H, Maruyama K, Muraki I, Tamakoshi A. Associations between dietary intakes of iron, copper and zinc with risk of type 2 diabetes mellitus: A large population-based prospective cohort study. Clin Nutr. 2018 Apr;37(2):667-674. doi: 10.1016/j.clnu.2017.02.010. Epub 2017 Feb 28. PMID 28285974
- [Background] Liamis G, Liberopoulos E, Barkas F, Elisaf M. Diabetes mellitus and electrolyte disorders. World J Clin Cases. 2014 Oct 16;2(10):488-96. doi: 10.12998/wjcc.v2.i10.488. PMID 25325058
- [Background] Hou Y, Xiang J, Dai H, Wang T, Li M, Lin H, Wang S, Xu Y, Lu J, Chen Y, Wang W, Ning G, Zhao Z, Bi Y, Xu M. New clusters of serum electrolytes aid in stratification of diabetes and metabolic risk. J Diabetes. 2022 Feb;14(2):121-133. doi: 10.1111/1753-0407.13244. Epub 2021 Dec 28. PMID 34963041
- [Background] Kieboom BCT, Ligthart S, Dehghan A, Kurstjens S, de Baaij JHF, Franco OH, Hofman A, Zietse R, Stricker BH, Hoorn EJ. Serum magnesium and the risk of prediabetes: a population-based cohort study. Diabetologia. 2017 May;60(5):843-853. doi: 10.1007/s00125-017-4224-4. Epub 2017 Feb 21. PMID 28224192
- [Background] Alvarez S, Coffey R, Mathias PM, Algotar AM. Prediabetes. 2023 Jul 17. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK459332/ PMID 29083606